CLINICAL TRIAL: NCT05983523
Title: A Phase I Study of PEP07 (Checkpoint Kinase 1 Inhibitor) in Patients with Advanced or Metastatic Solid Tumors
Brief Title: A Study of PEP07 (Checkpoint Kinase 1 Inhibitor) in Patients with Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaEngine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEP07-102
Record Dates: First submitted 2023-07-24; First posted 2023-08-09 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor
Keywords: Checkpoint Kinase 1 Inhibitor
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Masking Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PEP07 Monotherapy (Experimental): The dose escalation stage of PEP07 monotherapy consists of an accelerated dose escalation followed by a standard "3+3" dose escalation. The accelerated titration will enroll 1 patient in each dose cohort until 1 patient experiences a DLT or a total of 2 patients experience any ≥ grade 2 PEP07-related AE during Cycle 1, and then the dose escalation will be switched to the 3+3 scheme to enroll 3 to 6 patients at the dose cohort where the DLT or the second ≥ grade 2 PEP07-related AE is observed.
  To confirm the safety and evaluate the preliminary efficacy of PEP07, expansion cohorts with 12 patients will be opened for PEP07 monotherapy at RP2D once efficacy signal is observed in the dose escalation.
  Interventions: Drug: PEP07

INTERVENTIONS:
Drug: PEP07 — PEP07 is a potent, highly selective, orally bioavailable small molecule inhibitor of Chk1. PEP07 will be provided as 20 mg and 150 mg strength capsules to be administrated orally. Patients allocated to different dose levels of PEP07 monotherapy will receive either 20 mg or 150 mg oral capsules for 2 consecutive days followed by 5 days treatment off (2-on/5-off) schedule every week, 4 weeks as a treatment cycle.

SUMMARY:
The goal of this clinical trial is To establish the safety profile and determine the dose-limited toxicity (DLT) of PEP07 monotherapy in patients with advanced or metastatic solid tumors. To determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of PEP07 monotherapy.

Participants will receive PEP07 administered orally once daily (QD) for 2 consecutive days and 5 days off, every week for 4 weeks until disease progression, intolerable toxicity, confirmed pregnancy, death, consent withdrawal, or other anti-cancer treatment is required, or the Sponsor ends the study, whichever occurs first.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, multi-center study recruiting patients with advanced or metastatic solid tumors.

The study will utilize an Accelerated Titration Design in the lower dose levels followed by a traditional 3+3 dose escalation design at higher dose levels until RP2D is determined. The starting dose will be 40 mg.

All potential study candidates will provide informed consent and will undergo screening procedures before participating in the study. After a screening period of up to 28 days, qualified patients will be enrolled to receive their assigned dose regimen of PEP07 monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be ≥ 20 years of age

2a. For subject in the dose escalation stage: Subjects with advanced or metastatic solid tumors who have failed on or are intolerant to standard treatment or have no access to standard treatment.

2b. For subject in the dose expansion stage: Subjects with histologically or cytologically confirmed malignant solid tumors which are advanced or metastatic, who have failed on or are intolerant to standard treatment or have no access to standard treatment.

3. At least one measurable lesion according to the RECIST version 1.1.

4. Subjects must have ECOG Performance score of 0-1.

5. Subject must have adequate renal function as demonstrated by a calculated creatinine clearance ≥ 50 mL/min; determined via urine collection for 24-hour creatinine clearance or by the Cockcroft Gault formula.

6. Subject must have adequate liver function as demonstrated by:

* Aspartate aminotransferase (AST) ≤ 2.5 × ULN (≤ 5 × ULN, if attributable to liver metastases)
* Alanine aminotransferase (ALT) ≤ 2.5 × ULN (≤ 5 × ULN, if attributable to liver metastases)
* Bilirubin ≤ 1.5 × ULN

  7. Subject must have adequate bone marrow function as demonstrated by:
* Absolute neutrophil count (ANC) ≥ 1500/mm3
* Platelet counts ≥ 100,000/mm3
* Hemoglobin ≥ 9 g/dL

  8. Female subjects with reproductive potential must have a negative serum pregnancy test within 7 days prior to the first dose of study treatment. Women of childbearing potential as well as males of reproductive potential must agree to refrain from unprotected sex and ensure highly effective contraception with partner during study period and until 6 months after the last dose of study drug.

  9. Provision of signed and dated informed consent form.

Exclusion Criteria:

1. Pregnant or breastfeeding females.
2. Subjects have received anti-cancer therapy including chemotherapy, radiotherapy, hormonal or any investigational therapy within 14 days or 5 half-lives (whichever is shorter) or immunotherapy within 30 days prior to the first dose of study treatment.
3. Subjects have received strong or moderated cytochrome P450 3A4 (CYP3A4) inhibitors or CYP inducers such as ketoconazole, erythromycin, netupitant, isavuconazole etc. within 5 half-lives or 7 days (whichever is the shortest) prior to the first dose of study treatment.
4. Known history of or positive screening result for human immunodeficiency virus (HIV) antibody.
5. Viral hepatitis type B or C which require antiviral therapy, and/or have HBsAg (+) with HBV DNA ≥ 1000 IU/mL, or anti-HCV Ab (+) with HCV RNA (+). If a patient with HBsAg (+) then HBV DNA needs to be tested. If a patient with anti-HCV Ab (+) then the patient needs to be followed for HCV RNA (-) to be enrolled.
6. Uncontrolled systemic infection /or requiring isolation.
7. Patients with previous history of other malignant diseases within the last 5 years (other than adequately treated non-melanotic skin cancer, in-situ carcinoma of the uterine cervix or myelodysplastic syndromes).
8. Subjects with ongoing ≥ Grade 2 (CTCAE v5.0) toxicity (except alopecia and hot flashes) related to previous treatment.
9. Subjects have baseline QTcF interval > 450 msec at screening (within 28 days prior to the first dose of study treatment, mean of triplicate readings within approximately 5 minutes).
10. Subjects have cardiovascular disability status of New York Heart Association (NYHA) ≥ Class III, left ventricular ejection fraction < 45% at baseline, history of cardiac ischemia within the past 6 months, or prior history of cardiac arrhythmia requiring treatment.
11. Subjects have undergone any major surgery within 3 weeks prior to the first dose of study treatment.
12. Subjects with known active central nervous system (CNS) or leptomeningeal metastases. Subjects with previously-treated brain or meningeal metastases may participate and be eligible for treatment provided they are stable and asymptomatic (without evidence of progression by imaging of the brain at least 4 weeks prior to the first dose of study treatment), and are not using excessive steroids (defined as a prednisolone dose ≤ 10 mg daily or equivalent) for at least 2 weeks prior to the first dose of study treatment.
13. Subjects have had any of the following within 6 months prior to the first dose of study treatment: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or seizure disorder.
14. Subjects have any other medical or psychiatric condition that, in the opinion of the investigator, might interfere with the subject's participation in the trial or interfere with the interpretation of trial results.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2027-02-25 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
to find out the DLT | 4 weeks after first dosing
  To establish the safety profile and determinate the dose-limited toxicity (DLT) of PEP07 monotherapy
to find out the MTD and RP2D | 4 weeks after first dosing
  To determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of PEP07 monotherapy

SECONDARY OUTCOMES:
to know the PK profile | 6 months
  To assess the area under the plasma concentration versus time curve (AUC) of PEP07 as a monotherapy
to know the PK profile | 6 months
  To assess the time to maximun (peak) plasma concentration (Tmax) of PEP07 as a monotherapy
to know the PK profile | 6 months
  To assess the apparent half-life (t 1/2) of PEP07 as a monotherapy
to know the PK profile | 6 months
  To assess the peak plasma concentration (Cmax) of PEP07 as a monotherapy
to know the efficacy | from date of first dosing until the date of disease progressionfrom date of first dosing until the date of disease progression, assessed up to 12 months
  To assess the preliminary evidence of anti-tumor activities of PEP07 by objective response rate (ORR)
to know the efficacy | from date of first dosing until the date of disease progressionfrom date of first dosing until the date of disease progression, assessed up to 12 months
  To assess the preliminary evidence of anti-tumor activities of PEP07 by objective To assess the preliminary evidence of anti-tumor activities of PEP07 by progression free survival (PFS)
to know the efficacy | from date of first dosing until the date of disease progressionfrom date of first dosing until the date of disease progression, assessed up to 12 months
  To assess the preliminary evidence of anti-tumor activities of PEP07 by overall survival (OS)

OTHER OUTCOMES:
to find out the change in biomarkers | 6 months
  To assess Chk1 level in subjects with advanced or metastatic solid tumors
to find out the change in biomarkers | 6 months
  To assess γH2AX level in subjects with advanced or metastatic solid tumors
to find out the change in biomarkers | 6 months
  To assess pCHK1 level in subjects with advanced or metastatic solid tumors

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD